CLINICAL TRIAL: NCT04734613
Title: Tai Chi Applied Behavioral Modification Program for Individuals With Metabolic Syndrome: Randomized Study
Brief Title: Tai Chi for Behavioral Modification Among Individuals With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chungnam National University (Other)
Collaborators: National Research Foundation, Singapore (Other Government)
Responsible Party: Principal Investigator, Rhayun Song, Professor, Chungnam National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ChungnamNU2
Record Dates: First submitted 2021-01-26; First posted 2021-02-02 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Aquatic Therapy; Self-Management

STUDY DESIGN:
Intervention Model Description: randomized trial to assign the participants either to intervention group 1 (Tai Chi exercise) or to intervention group 2 (self management)
Who Masked: Outcomes Assessor
Masking Description: blood sample will be analyzed by the lab technician without identity of the group assignment. self-reported questionnaire is also used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai Chi intervention (Experimental): Tai Chi exercise intervention provided twice a week for one hour for 12 weeks
  Interventions: Behavioral: Tai Chi exercise
- self management (Active Comparator): self management program provided 6 sessions (one hour per session) for 12 weeks
  Interventions: Behavioral: self management

INTERVENTIONS:
Behavioral: Tai Chi exercise — Yang style Tai Chi 16 movements
  Arms: Tai Chi intervention
Behavioral: self management — health education and dietary counseling
  Arms: self management

SUMMARY:
This is the randomized trial to explore the effect of behavioral modification program (Tai Chi vs. self management) on adults with metabolic syndrome. The outcome variables include health behavior, metabolic syndrome indicators, quality of life.

DETAILED DESCRIPTION:
1. venue: the individuals with diagnosis of metabolic syndrome are recruiting from university hospital outpatient clinic or primary clinic.
2. inclusion criteria: diagnosed of metabolic syndrome, agree to participate either programs, no history of participating regular exercise program past 6 months.
3. intervention: The behavioral modification program consisting of Tai Chi exercise (twice a week for 12 weeks) and self-management program (6 sessions every two weeks) is provided to the participants who randomly assigned to either group. Short form Yang style Tai Chi (16 movements) were led by trained Tai Chi practitioners, and self-management program were provided by nurse educators.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of metabolic syndrome
* adults who agree to participate either behavioral modification programs for 12 weeks
* be able to understand the questionnaire and follow the exercise or education program

Exclusion Criteria:

* who attend regular exercise program past 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Change in Cardiac health behavior scale | change from baseline health behavior score at 3 months
  cardiac health behaviors scale including exercise, diet, stress management, health responsibility, and smoking - 25 items in 4 point Likert scale
Change in blood pressure | change from baseline blood pressure at 3 months
  systolic and diastolic blood pressure (mmHg)
change in lipid profile | change from baseline lipid profile at 3 months
  high density lipoprotein(HDL), low density lipoprotein(LDL), total cholesterol, triglyceride
Change in blood glucose | change from baseline blood glucose at 3 months
  HbA1C
Change in abdominal obesity | change from baseline waist circumference at 3 months
  waist circumference (in centimeters) will be measured with indicator on upper hip bone

SECONDARY OUTCOMES:
Change in quality of life | change from baseline QOL score at 3 months
  health related quality of life (by SF36 v.2) to calculate mental and physical components in 100 points

CONTACTS AND LOCATIONS:
Overall Officials: Rhayun Song, Principal Investigator — Chungnam National University
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea